CLINICAL TRIAL: NCT01902602
Title: Grand Autohemo-Therapy With Oxygen-ozone on Patients With Hypertonia
Acronym: HAB
Status: Terminated | Type: Observational
Why Stopped: Lack of compliance of the clinical site
Sponsor: Herrmann Apparatebau GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: HAB10-2012
Record Dates: First submitted 2013-07-15; First posted 2013-07-18 (Estimated); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Hypertonia
MeSH Terms: conditions — Muscle Hypertonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this clinical study is to evaluate the influence of the Great autohemotherapy with oxygen-ozone (hyperbaric ozone therapy ) to describe the cardiovascular system in patients with resistant hypertension. The primary endpoint is the change in mean blood pressure after 10 treatments .

In addition, data are collected on the immune system as well as for food and sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* Resistant Hypertension > 140 / > 90mmHg
* Inclusion age : 45 +
* Regular monitoring of blood levels considered
* pre-medication to lower blood pressure for at least 3 weeks before the preliminary investigation consistent
* Men and Women

Exclusion Criteria:

* derailed diabetes
* renal impairment , renal creatinine clear <50 ml
* Non - austherapierte cancer / tumor patients
* Non - adjusted thyroid dysfunction
* BMI> 35
* LVEF <limit ( " 35% " )
* Peripheral AVK ( ABI - measurement ) > Stage II
* regurgitation > Stage I
* abdominal aneurysm
* infections
* acute febrile infections with temperature > 38.5 ° C
* COPD and asthma to stage III
* dyspnea NYHA > Stage III
* z.n. Stroke shorter than 12 weeks
* Acute liver failure
* Acute Apoplexy
* Severe poisoning
* drug addiction
* hyperthyroidism
* Hypotension
* hypocalcemia
* hypoglycemia
* ozone allergy
* pregnancy
* clotting problems ( hemophilia )
* pre-existing condition with hemoglobin < 9mg/dl
* Fresh myocardial infarction
* Internal bleeding
* thrombocytopenia
* Acute alcohol
* Citrus allergy when using sodium citrate

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients which fulfill the mentioned criterias.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change of blood pressure | 3 months
  Primary endpoint is, that there is a changing of the middle blood pressure after 10 treatments. The blood pressure will get messured at all patients which get treated with oxygen-ozone. The aim is reached, if there is a reduction of the middle blood pressure after 10 treatments by 10 mmHg compared to the blood pressure by the patients at the baseline at beginning.

SECONDARY OUTCOMES:
Change of pulse | 3 months
  The Pulse will be measured at each follow-up. It will be measured 3 times at the dominate arm.
Change of blood count, liver and nephrew values | 3 months
  The change of blood counts, liver and nephrew values serves as a sign for change of immune activity in a patient. Furthermore potential negative effects will be reportet as an adverse event.
Change of liver and nephrew values | 3 months
Change of life and Sleeping quality | 3 months
  Change of life and sleeping quality will be measured in a 7 scale. This questionnaire is to fill in by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Panos Porikis, Phd, Principal Investigator — unafflicated
Locations (1):
- Dr. Panos Porikis, Biblis, Hesse, Germany